CLINICAL TRIAL: NCT02822066
Title: Effectivity and Safety of Irreversible Electroporation for Refractory Neoplasms in Liver and Pancreas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA-003
Record Dates: First submitted 2016-06-20; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Refractory Neoplasms
Keywords: Effectivity; safety; irreversible electroporation; liver; pancreas
MeSH Terms: conditions — Neoplasms | interventions — Electroporation

ARMS (1):
- IRE for refractory neoplasms in liver and pancreas (Experimental): To evaluate the safety and efficacy of irreversible electroporation (IRE) for refractory neoplasms in liver and pancreas, the investigators used preoperative and postoperative US/CEUS/CT/MRI to assess lesions, and laboratory tests including the tumor markers to evaluate the general condition of patients. Intraoperative US/CEUS/CT would be applied to monitor ablation lesions.
  Interventions: Procedure: Electroporation

INTERVENTIONS:
Procedure: Electroporation — Effectivity and safety of irreversible electroporation for refractory neoplasms in liver and pancreas

SUMMARY:
The pupose of this study is to evaluate the safety and efficacy of irreversible electroporation (IRE) for refractory neoplasms in liver and pancreas, the investigators used preoperative and postoperative US/CEUS/CT/MRI to assess lesions, and laboratory tests including the tumor markers to evaluate the general condition of patients. Intraoperative US/CEUS/CT would be applied to monitor ablation lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hepatic portal focal lesion adjacent to important structures like bile duct and portal blood vessels, or intolerant surgery.
2. Patients with pancreatic cancer adjacent to blood vessels, or intolerant surgery.

Exclusion Criteria:

Patients with:

1. Metal in the body
2. ChildPugh ≥ 3
3. Long-term use of anticoagulant drugs including warfarin, clopidogrel bisulfate
4. Poor cardiac or renal function with intolerant surgery or anesthesia.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
60 patients of refractory neoplasms in liver and pancreas with irreversible electroporation-related effectivity as assessed by MRI | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Dollinger M, Zeman F, Niessen C, Lang SA, Beyer LP, Muller M, Stroszczynski C, Wiggermann P. Bile Duct Injury after Irreversible Electroporation of Hepatic Malignancies: Evaluation of MR Imaging Findings and Laboratory Values. J Vasc Interv Radiol. 2016 Jan;27(1):96-103. doi: 10.1016/j.jvir.2015.10.002. PMID 26777402
- [Result] Froud T, Venkat SR, Barbery KJ, Gunjan A, Narayanan G. Liver Function Tests Following Irreversible Electroporation of Liver Tumors: Experience in 174 Procedures. Tech Vasc Interv Radiol. 2015 Sep;18(3):140-6. doi: 10.1053/j.tvir.2015.06.004. Epub 2015 Jun 18. PMID 26365543
- [Result] Hosein PJ, Echenique A, Loaiza-Bonilla A, Froud T, Barbery K, Rocha Lima CM, Yrizarry JM, Narayanan G. Percutaneous irreversible electroporation for the treatment of colorectal cancer liver metastases with a proposal for a new response evaluation system. J Vasc Interv Radiol. 2014 Aug;25(8):1233-1239.e2. doi: 10.1016/j.jvir.2014.04.007. Epub 2014 May 24. PMID 24861662
- [Result] Belfiore MP, Ronza FM, Romano F, Ianniello GP, De Lucia G, Gallo C, Marsicano C, Di Gennaro TL, Belfiore G. Percutaneous CT-guided irreversible electroporation followed by chemotherapy as a novel neoadjuvant protocol in locally advanced pancreatic cancer: Our preliminary experience. Int J Surg. 2015 Sep;21 Suppl 1:S34-9. doi: 10.1016/j.ijsu.2015.06.049. Epub 2015 Jun 25. PMID 26118600
- [Result] Lambert L, Horejs J, Krska Z, Hoskovec D, Petruzelka L, Krechler T, Kriz P, Briza J. Treatment of locally advanced pancreatic cancer by percutaneous and intraoperative irreversible electroporation: general hospital cancer center experience. Neoplasma. 2016;63(2):269-73. doi: 10.4149/213_150611N326. PMID 26774149
- [Result] Paiella S, Butturini G, Frigerio I, Salvia R, Armatura G, Bacchion M, Fontana M, D'Onofrio M, Martone E, Bassi C. Safety and feasibility of Irreversible Electroporation (IRE) in patients with locally advanced pancreatic cancer: results of a prospective study. Dig Surg. 2015;32(2):90-7. doi: 10.1159/000375323. Epub 2015 Feb 28. PMID 25765775
- [Derived] Jiang T, Zhao Q, Tian G, Chen X, Wu L. Irreversible electroporation ablation of end-stage metastatic retroperitoneal lesions: Report on three cases and literature review. Exp Ther Med. 2019 Sep;18(3):2243-2249. doi: 10.3892/etm.2019.7780. Epub 2019 Jul 17. PMID 31410175